CLINICAL TRIAL: NCT05018338
Title: Pre-pilot Study of Brain-Shift Monitoring Using 3D Scanning
Brief Title: Brain-Shift Monitoring Using 3D Scanning
Status: Terminated | Type: Observational
Why Stopped: Low enrollment of subjects
Sponsor: Advanced Scanners Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 0100
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Craniotomy for Epilepsy and Malignant Tumor Removal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- The study cohort: The study will enroll 10 subjects meeting the eligibility criteria, with the expectation to obtain complete data from at least 6 subjects.
  Interventions: Device: Brain shift monitoring

INTERVENTIONS:
Device: Brain shift monitoring — For use to monitor brain shift during craniotomy
  Other Names: 3D brain scanning

SUMMARY:
A prospective non-invasive data/image collection for evaluation of the performance of the Advanced Scanners 3D scanner during brain surgery.

The primary objective is to evaluate the performance of the scanner in determining the brain surface shape over multiple time points during craniotomies (surgical opening into the skull), and present those shapes in full color, with high resolution in all three coordinates of 3D space. A secondary objective is to use the measurements to determine brain shift as a function of time.

DETAILED DESCRIPTION:
The scanner sterilization will largely follow procedures used currently for cameras and microscopes: the scanner will be draped in a disposable drape custom manufactured for the device by a leading instrument drape manufacturer (Medline). The drape will be windowed with a sterilized shatterproof plastic optical window. Standard hospital procedures will be followed for the disposal of instrument drapes. The drape will be sterile and wrapped in the conventional manner, and the drape itself will be disposable. Prior to surgery, the drape, window and frame will undergo the same sterilization procedure as other equipment. If window transparency is compromised during surgery, it can be cleaned with a cleaning agent.

The scanner will illuminate the craniotomy region with light for the duration of its use, which may be for the duration of the surgery. The scanner will be anywhere from 8 to 12 inches away from the patient, illuminating the subject's brain by the scanner light for 2 minutes at a time, or continuously, either with or without maximum overhead lighting.

For each patient, the duration of obtaining data will last for the duration of the clinical operation procedure. The 3D Scanner on and off time would add less than 5 minutes to the procedure, not including measurement time.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 6 years of age at Visit 1.
2. Clinically planned for craniotomy, including for malignant tumors, whether awake or under general anesthesia.
3. Able to provide written informed consent (and assent when applicable) - by subject or subject's legal representative - and agrees to comply with the requirements of the study.

Exclusion Criteria:

1. Language problems that would prevent from properly understanding instructions.
2. Requirement of an interpreter.
3. Patients who are excluded from consideration for the clinical operation are therefore excluded from the research study.
4. Special populations: pregnant women, prisoners.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects seen by Dr. Anat I. Patel (neurosurgeon) and scheduled for craniotomy at St. David's North Austin Medical Center are the potential population for this study.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Brain-shift measurement | Throughout the surgical procedure
  Measure brain-shift in human subjects' brains with our scanning technology, and compare with preoperative MRI or CT, and, optionally, with inter-operative or postoperative MRI or CT scans. Measurements will include changes, measured in millimeters, of the surface anatomic features of the brain from the optical scans. Overall topological changes will also be measured between pre- and post-operative CT/MRI imaging of the patient with the optical scans. All these measurements will be performed using co-registered surfaces, reporting specifically computer-determined measurement of distances between those surfaces.

SECONDARY OUTCOMES:
Brain-shift measurement accuracy | Throughout the surgical procedure
  Measurement of brain-shift in human subjects' brains with sub-mm accuracy using our scanning technology

OTHER OUTCOMES:
Operation of the 3D scanner | Throughout the surgical procedure
  Successful operation of the scanner providing periodic feedback to the surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Bernstein, PhD, Study Director — Advanced Scanners Inc.
Locations (1):
- St. David's Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
If data is shared, it will be anonymized.

REFERENCES:
- [Background] Daanen, H. A. M. & Ter Haar, F. B. 3D whole body scanners revisited. Displays 34, 270-275 (2013).
- [Background] Yang, J. C. et al., Journal of Clinical Neuroscience 21, p. 1230 (2014) and Mert, A. et al, Operative Neurosurgery 71, p. 286 (2012), respectively.
- [Background] Zhang, D., Lu, G., Li, W., Zhang, L. & Luo, N. Palmprint Recognition Using 3-D Information. IEEE Transactions on Systems, Man, and Cybernetics, Part C (Applications and Reviews) 39, 505-519 (2009).
- [Background] Park HK, Chung JW, Kho HS. Use of hand-held laser scanning in the assessment of craniometry. Forensic Sci Int. 2006 Jul 13;160(2-3):200-6. doi: 10.1016/j.forsciint.2005.10.007. Epub 2005 Nov 9. PMID 16289612
- [Background] Kovacs L, Zimmermann A, Brockmann G, Guhring M, Baurecht H, Papadopulos NA, Schwenzer-Zimmerer K, Sader R, Biemer E, Zeilhofer HF. Three-dimensional recording of the human face with a 3D laser scanner. J Plast Reconstr Aesthet Surg. 2006;59(11):1193-202. doi: 10.1016/j.bjps.2005.10.025. Epub 2006 Mar 9. PMID 17046629
- [Background] Hameeteman M, Verhulst AC, Vreeken RD, Maal TJ, Ulrich DJ. 3D stereophotogrammetry in upper-extremity lymphedema: An accurate diagnostic method. J Plast Reconstr Aesthet Surg. 2016 Feb;69(2):241-7. doi: 10.1016/j.bjps.2015.10.011. Epub 2015 Oct 22. PMID 26590631
- [Background] Arlt F, Chalopin C, Muns A, Meixensberger J, Lindner D. Intraoperative 3D contrast-enhanced ultrasound (CEUS): a prospective study of 50 patients with brain tumours. Acta Neurochir (Wien). 2016 Apr;158(4):685-694. doi: 10.1007/s00701-016-2738-z. Epub 2016 Feb 16. PMID 26883549